CLINICAL TRIAL: NCT04797234
Title: Evaluation of the Effects of Roper, Logan and Tierney Nursing Model Based Patient Education Program on the Daily Living Activities and Self-Care Power of Hemodialysis Patients
Brief Title: The Effect of Patient Education Based on Nursing Model on Life Activities and Self-Care of Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 10879717-050.01.04
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Hemodialysis Complication
Keywords: education; hemodialysis; life model; self-care

STUDY DESIGN:
Intervention Model Description: The research is carried out to evaluate the effects of the education given to individuals who receive hemodialysis treatment based on Roper, Logan - Tierney's Nursing Model on the independence level and self-care power of the sick individuals in their daily living activities. The research is planned to be conducted as a randomized controlled study determined by simple random method, two groups, pretest - posttest, and experimental research design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): There will be no intervention to the control group.
  Interventions: Other: Control
- Experiment (Experimental): The experimental group will be trained for 6 weeks.
  Interventions: Other: Experiment

INTERVENTIONS:
Other: Control — There will be no intervention to the control group.
  Arms: Control
Other: Experiment — The experimental group will be trained for 6 weeks.
  Arms: Experiment

SUMMARY:
Chronic Renal Failure (CRF); The result of a decrease in the glomerular filtration value is defined as a chronic and progressive deterioration in the fluid-solute balance of the kidney and metabolic-endocrine functions. Treatment is kidney transplant or dialysis. CRF affects 10-15% of adults worldwide. CRF rate in the general adult population in Turkey is 15.7%. According to the data of the Turkish Nephrology Association, renal replacement therapy (RRT) is applied to a total of 77,311 patients in our country by the end of 2017. The most common (76%) applied RRT type is hemodialysis treatment. In individuals receiving hemodialysis treatment, nausea-vomiting, weakness, fatigue, itching, fluid-solute imbalances, hypotension and pain can be seen due to uremia. This situation reduces the functionality of the patient and the limitation of physical activities brings physical and psycho-social effects with it. The dependence of the individual on the dialysis machine, the healthcare team and the family in treatment programs that last three days a week, on average four hours a day, affects the personal lives of the patients. It can be said that nursing care and education are of great importance in resolving the existing or potential problems of patients who are dependent on hemodialysis as a result of CRF, and in adapting patients to life with their disease. It is the nursing theories that will guide these attempts of nurses. Because nursing theories interpret and define the profession; thus helping nurses in training, practice and research activities as a professional. Nursing Model of Roper, Logan-Tierney (RLT), one of the important theories of nursing, is based on the life model. In this model, the main purpose of nursing is to ensure that people are informed so that they can lead a quality and healthy life. This model, which can be integrated into all service areas of the health care system and handles individual-centered care with a humanistic and holistic approach, supports the participation of the individual in care. It is predicted that the patient education program created using the Nursing Model of RLT will support the increase of the independence levels and self-care abilities of individuals who receive hemodialysis treatment.

DETAILED DESCRIPTION:
Chronic Renal Failure (CRF); The result of a decrease in the glomerular filtration value is defined as a chronic and progressive deterioration in the fluid-solute balance of the kidney and metabolic-endocrine functions. CRF is an irreversible, progressive disease involving many systems. Its treatment is kidney transplant or dialysis. CRF affects 10-15% of adults worldwide. In other words, one out of every six adults has CRF. CRF rate in the general adult population in Turkey is 15.7%. According to the data of the Turkish Nephrology Association, renal replacement therapy (RRT) is applied to a total of 77,311 patients in our country as of the end of 2017. The most common (76%) applied RRT type is hemodialysis treatment. In individuals receiving hemodialysis treatment, nausea-vomiting, weakness, fatigue, itching, fluid-solute imbalances, hypotension and pain can be seen due to uremia. This situation reduces the functionality of the patient and the limitation of physical activities brings physical and psycho-social effects with it. The dependence of the person on the dialysis machine, the healthcare team and the family in the treatment programs that last three days a week, an average of four hours a day, affects the personal lives of the patients. It can be said that nursing care and education are of great importance in resolving the existing or potential problems of patients whose CRF result is due to hemodialysis, and in adapting patients to life with their disease. It is the nursing theories that will guide these attempts of nurses. Because nursing theories interpret and define the profession; thus helping nurses in training, practice, research activities as a professional. Nursing Model of Roper, Logan-Tierney (RLT), one of the important theories of nursing, is based on the life model. In this model, the main purpose of nursing is to ensure that people are informed so that they can lead a quality and healthy life. In the "Nursing Model" developed by RLT based on the Life Model, they focused on providing nursing care based on human characteristics, believed in the necessity of observations and measurable events and activities, and based their nursing services on these beliefs. This model, which can be integrated into all service areas of the health care system and handles individual-centered care with a humanistic and holistic approach, supports the participation of the individual in care. It is predicted that the patient education program created using the Nursing Model of RLT will support the increase of the independence levels and self-care abilities of individuals who receive hemodialysis treatment. In this study, it is planned to evaluate the effect of the education given to individuals receiving hemodialysis based on Roper, Logan-Tierney's Nursing Model on the level of independence and self-care ability in daily living activities.

Research for the development of the nursing profession contributes to the knowledge of nursing science by developing and testing nursing models / theories. In the literature, it is seen that the use of the Nursing Model of RLT is limited only by mentioning the content of the theory in certain parts of the study rather than reflecting it on the whole study. There are no extensive explanations about the model and enough information about how it can be used in practice. It has been determined that postgraduate studies conducted using the Nursing Model of RLT are mostly descriptive studies. However, nursing theories and models should be used effectively in research and practice. When the studies on individuals who receive hemodialysis treatment are examined, it has been determined that the use of the Nursing Model of RLT is very low. It is predicted that the patient education program created using this Nursing Model will support the increase of the independence levels and self-care abilities of individuals who receive hemodialysis treatment.

At the end of the patient education program based on the Nursing Model of RLT, individuals who receive hemodialysis treatment will increase their independence levels and self-care abilities in daily living activities. It will be ensured that caregiving healthcare professionals perform hemodialysis treatment with less stress.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and over, who agree to participate in the research, Receiving hemodialysis for 4 hours 3 days a week,
* Having received hemodialysis treatment for at least 1 year and continuing the treatment,
* Without cognitive, affective and mental limitations,
* It will create all hemodialysis patients who do not have a communication problem regarding vision and hearing.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-02-06 (Actual); Study Completion 2021-05-08 (Actual)

PRIMARY OUTCOMES:
Self-Care Ability Scale | 6 weeks
  It is a scale used to measure an individual's self-care ability or self-care ability. The maximum score is 140. The higher the score obtained from the scale indicates the high level of self-care or self-care ability and power of the individual.

SECONDARY OUTCOMES:
Modified Barthel Index | 6 weeks
  The Modified Barthel Index is a comprehensive scale that can be used to measure patients' physical abilities. The total score that can be obtained from the Modified Barthel Index is between 0 and 100, with 0 points showing full dependency and 100 points showing full independence.

CONTACTS AND LOCATIONS:
Overall Officials: Abdulsamed Kaya, Principal Investigator — MUS ALPARLAN UNIVERSITY
Locations (1):
- Mus Alparlan University, Muş, Turkey (Türkiye)